CLINICAL TRIAL: NCT07132216
Title: Effect of Virtual Reality on Intraoperative Anxiety, Stress and Patient's Satisfaction Among Palestinian Patients Undergoing Regional Anesthesia
Brief Title: Effect of Virtual Reality on Anxiety, Stress, and Patient's Satisfaction Among Patients Undergoing Regional Anesthesia
Acronym: VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, khulud "Mohammad Hasham" Hasham Mansor, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB RHDIRB2019041701
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Perioperative Anxiety; Perioperative Stress; Patient Satisfaction; Regional Anesthesia; Elective Surgery
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Participants in the VR group received immersive VR intervention during the operation using head-mounted devices, while the control group received routine care.
  The Meta Quest 2 VR headset with built-in headphones was used. Patients selected VR environments from a predefined list of five nature scenes (beach, forest, mountain, underwater, and meadow) with identical meditation audio tracks lasting 30 minutes each.
  Guided Meditation VR from Cubicle Ninjas featured 360-degree nature environments with standardized calming background music and guided meditation narration. VR was applied immediately after spinal anesthesia before the surgical incision. Sessions lasted 30 minutes and were discontinued if the patient reported nausea, dizziness, or requested removal.
Masking Description: Patients were not blinded due to the VR intervention, but the anesthesiologist and outcome assessors were blinded to group assignments. To maintain blinding for the anesthesiologist, VR headsets were covered with opaque drapes during clinical assessments, and research staff members not involved in clinical care managed the VR equipment. The anesthesiologist was only informed of group allocation after completing all clinical assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes

ARMS (2):
- VR group (Experimental): The Meta Quest 2 VR headset with built-in headphones was used. Patients selected VR environments from a predefined list of five nature scenes (beach, forest, mountain, underwater, and meadow) with identical meditation audio tracks lasting 30 minutes each. Guided Meditation VR from Cubicle Ninjas (https://guidedmeditationvr.com/)featured 360-degree nature environments with standardized calming background music and guided meditation narration. VR was applied immediately after spinal anesthesia and before the surgical incision. Sessions lasted 30 minutes and were discontinued if the patient reported nausea, dizziness, or requested removal.
  Interventions: Device: Meta Quest 2 VR headset
- control group (No Intervention): Participants in the control group only receive standard care according to the hospital's protocol during the operation.

INTERVENTIONS:
Device: Meta Quest 2 VR headset — The Meta Quest 2 VR headset with built-in headphones was used. Patients selected VR environments from a predefined list of five nature scenes (beach, forest, mountain, underwater, and meadow) with identical meditation audio tracks lasting 30 minutes each. Guided Meditation VR from Cubicle Ninjas (https://guidedmeditationvr.com/)featured 360-degree nature environments with standardized calming background music and guided meditation narration. VR was applied immediately after spinal anesthesia and before the surgical incision. Sessions lasted 30 minutes and were discontinued if the patient reported nausea, dizziness, or requested removal.
  Arms: VR group

SUMMARY:
The goal of this clinical trial was to investigate the effect of Virtual Reality (VR) on intraoperative anxiety, stress, and patient satisfaction among Palestinian patients undergoing regional anesthesia. The study aimed to determine the efficacy and safety of VR as a non-pharmacological intervention during surgery. The main research hypotheses are:

H0: There will be no significant difference in anxiety levels between patients who receive immersive VR during regional anesthesia and those who do not receive pre- and post-virtual reality therapy.

H0: There will be no significant difference in perceived stress levels between patients who receive immersive VR during regional anesthesia and those who do not receive pre- and post-virtual reality therapy.

H0: There will be no significant difference in satisfaction levels between patients who receive immersive VR during regional anesthesia and those who do not receive pre- and post-virtual reality therapy.

Participants will:

Receive either VR intervention or standard care during their surgery. Complete assessments of anxiety and stress before and after the procedure using validated scales.

Provide feedback on their satisfaction levels post-operation using a Visual Analog Scale.

Be monitored for hemodynamic parameters throughout the surgical process.

DETAILED DESCRIPTION:
Title: Effect of Virtual Reality on Intraoperative Anxiety, Stress, and Patient Satisfaction among Palestinian Patients Undergoing Regional Anesthesia

Background: Preoperative and intraoperative anxiety and stress are common psychological responses that negatively impact surgical outcomes and patient satisfaction. While pharmacological interventions are traditionally used to manage these responses, non-pharmacological methods such as virtual reality (VR) are gaining prominence. This study aimed to evaluate the effect of VR on intraoperative anxiety, stress, and patient satisfaction among Palestinian patients undergoing regional anesthesia.

Methods: A randomized controlled trial was conducted at Rafidia Governmental Surgical Hospital in Nablus, Palestine, from June to September 2024. A total of 150 patients scheduled for elective urological surgery under regional anesthesia were randomly assigned into VR (n=75) and control (n=75) groups. Participants in the VR group received immersive VR intervention during the operation using head-mounted devices, while the control group received routine care. Anxiety was assessed using the State-Trait Anxiety Inventory (STAI), stress using the Perceived Stress Scale (PSS-10), and patient satisfaction using the Visual Analog Scale (VAS). Hemodynamic parameters were also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective urological surgery under regional anesthesia
* Patients older than 18 years
* Patients with no history of previous surgeries
* Patients suffering from moderate to severe anxiety and stress

Exclusion Criteria:

* Patients with a history of psychiatric disorders, epilepsy, hypertension, or chronic pain
* Patients who are mute and cannot read or write; patients with visual, hearing, or cognitive impairment
* Patients with implanted hearing aids or cardiac pacemakers
* Patients who received any anxiolytic, sedative, or hypnotic drugs before or during regional anesthesia
* Patients exposed to anesthetic or surgical complications during the operation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory (STAI) | preoperative and then 60 minutes postoperatively
  The STAI score ranges between 20-80, the higher score indicating greater anxiety. It is classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
Perceived Stress Scale (PSS-10) | preoperative and 60 minutes postoperatively
  The PSS-10 score can range from 0 to 40 with higher scores indicating higher perceived stress. It is classified as "no or low anxiety" (0-13), "moderate anxiety" (14-26), and "high anxiety" (27-40).

CONTACTS AND LOCATIONS:
Locations (1):
- Rafidia Surgical Governmental Hospital, Nablus City, West Bank, Palestine, Nablus, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No
This research was conducted to achieve a PhD degree.The paper is currently under review for publication, and sharing it before the review process is complete could violate journal policies.

REFERENCES:
- [Derived] Mansor K, Abdellatif SA, Mohamed NA. Virtual reality for reducing intraoperative anxiety and improving patient satisfaction under regional anesthesia among palestinian patients: a randomized controlled trial. BMC Anesthesiol. 2025 Nov 27;25(1):593. doi: 10.1186/s12871-025-03475-3. PMID 41310456
- See also: the website Guided Meditation VR application, developed by Cubicle Ninjas Agency — https://guidedmeditationvr.com/